CLINICAL TRIAL: NCT00115440
Title: BPA-Mediated Boron Neutron Capture Therapy (BNCT) in the Treatment of Glioblastoma or Anaplastic Astrocytoma Progressing After Conventional External Beam Radiotherapy
Brief Title: BNCT to Treat Glioma That Has Progressed Following Radiotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boneca Corporation (Industry)
Responsible Party: Markku Pohjola, Boneca Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIN-BNCT-03/2000; BNCT P-03
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2007-09

CONDITIONS: Glioblastoma; Anaplastic Astrocytoma
Keywords: glioblastoma; anaplastic astrocytoma; boron neutron capture therapy; radiation therapy; boronophenylalanine
MeSH Terms: conditions — Glioblastoma; Astrocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Active treatment arm.
  Interventions: Radiation: Bononophenylalanine (BPA)-based BNCT

INTERVENTIONS:
Radiation: Bononophenylalanine (BPA)-based BNCT — Boronophenylalanine is infused into a peripheral vein prior to neutron irradiation.

SUMMARY:
Boron Neutron Capture Therapy (BNCT) is an experimental radiation therapy technique which is based on the principle of irradiating boron atoms with neutrons. When neutrons have relatively low energy, boron atoms that have been targeted to cancerous tissue using a suitable boron carrier (an amino acid derivative called BPA, boronophenylalanine) will capture the neutrons. As a result from the neutron capture the boron atoms will split into two, producing helium and lithium ions. The helium and lithium ions, in turn, have only a short pathlength in tissue (about 5 micrometers) and will deposit their cell damaging effect mainly within the tumor provided that the boron carrier (BPA) has accumulated in the tumor. In practice, the study participants will receive BPA as an approximately 2-hour intravenous infusion, following which the tumor is irradiated with low energy (epithermal) neutrons obtained from a nuclear reactor at the BNCT facility. BNCT requires careful radiation dose planning, but neutron irradiation will last approximately only for one hour. In this study BNCT is given once. The study hypothesis is that anaplastic astrocytomas and glioblastomas that have recurred following conventional radiotherapy might accumulate the boron carrier compound, and might respond to BNCT.

DETAILED DESCRIPTION:
This is a single BNCT-facility, non-randomized, non-comparative, prospective, open-label, phase I/II study to determine the value of BNCT in the treatment of inoperable, irradiated, progressing anaplastic astrocytomas or glioblastomas following conventional radiation therapy. The neutron irradiation site is the FiR 1 reactor site, located at Otaniemi, Espoo, Finland, about 6 kilometers from the Helsinki University Central Hospital, Helsinki, where patient evaluation and post-irradiation care will take place.

BPA is infused as a fructose complex (BPA-F) into a peripheral vein over 2 hours prior to neutron irradiation. Blood samples will be taken before starting the BPA infusion, and thereafter at 20 to 40 minute intervals during the infusion, following infusion, and after delivering neutron irradiation to monitor the blood boron concentration. The blood samples will be analyzed for boron to estimate the average blood boron level during neutron irradiation. A minimum tumor dose of 17 Gy (W) is given while limiting the normal brain maximum peak dose to 8 Gy (W), and the average normal brain dose to 6 Gy (W). The first 10 patients will be given BPA 290 mg/kg, following which the BPA dose will be escalated in cohorts of 3 subjects gradually up to 450 mg/kg, provided that protocol-specified unacceptable toxicity will not occur.

All patients will be evaluated for response using CT or magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed supratentorial glioblastoma or anaplastic astrocytoma.
* Recurred tumor after surgery and radiotherapy or tumor progressing after radiotherapy.
* Recurrence/progression has been confirmed by serial MRI scans and a biopsy, or by debulking surgery.
* The World Health Organization performance status <2.
* WBC >2,500/mm3, platelet count >75,000/mm3, serum creatinine <180 umol/L.
* A written informed consent

Exclusion Criteria:

* Age less than 18
* Tumor infiltrates into the brain stem or the optic tracts
* The majority of tumor tissue consists of grade II glioma with only a focal grade III component
* A minimum gross tumor dose of 17 Gy (W) is not obtained in dose-planning
* Less than 6 months has elapsed from the last date of external irradiation
* Less than 4 weeks has elapsed from the last cancer chemotherapy dose prior to giving BNCT
* The total conventional radiation therapy dose given is more than 61 Gy or less than 50 Gy, or one of nonconventional fractionation schemes has been used (conventional: 1.8-2.0 Gy/day, 5 days per week, weekly dose 9 to 10 Gy)
* More than approximately 1/3 of the total brain volume has been within the 90% isodose
* Gliomas where the enhancing tumor volume is larger than 2/3 of the volume of one hemisphere in the MRI examination preceding BNCT
* More than one radiotherapy course has been given to the brain tumor
* Untreated congestive heart failure or renal failure
* Uncontrolled brain oedema despite the use of corticosteroids
* A cardiac pace-maker or an unremovable metal implant present in the head and neck region that will interfere with MRI-based dose-planning
* Restlessness or inability to lie in a cast for 30 to 60 minutes
* Clinical follow-up after therapy cannot be arranged
* Pregnancy
* Inability to understand treatment options
* Unwillingness to take part in the follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2001-03; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
safety | 3 years

SECONDARY OUTCOMES:
survival | 3 years
adverse effects of BNCT | 3 years
quality-of-life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Heikki T Joensuu, M.D., prof., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Department of Oncology, Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Background] Kouri M, Kankaanranta L, Seppala T, Tervo L, Rasilainen M, Minn H, Eskola O, Vahatalo J, Paetau A, Savolainen S, Auterinen I, Jaaskelainen J, Joensuu H. Undifferentiated sinonasal carcinoma may respond to single-fraction boron neutron capture therapy. Radiother Oncol. 2004 Jul;72(1):83-5. doi: 10.1016/j.radonc.2004.03.016. PMID 15236879
- [Result] Joensuu H, Kankaanranta L, Seppala T, Auterinen I, Kallio M, Kulvik M, Laakso J, Vahatalo J, Kortesniemi M, Kotiluoto P, Seren T, Karila J, Brander A, Jarviluoma E, Ryynanen P, Paetau A, Ruokonen I, Minn H, Tenhunen M, Jaaskelainen J, Farkkila M, Savolainen S. Boron neutron capture therapy of brain tumors: clinical trials at the finnish facility using boronophenylalanine. J Neurooncol. 2003 Mar-Apr;62(1-2):123-34. doi: 10.1007/BF02699939. PMID 12749708